CLINICAL TRIAL: NCT01943279
Title: A Comparison of Remote Follow-up After Medical Abortion Using Telephone and Serum Pregnancy Testing With Standard In-person Follow-up
Brief Title: Comparison of Telephone Follow-up With In-person Follow-up After Medical Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Responsible Party: Principal Investigator, Sheila Dunn, MD, MSc, CCFP(EM), FCFP, Women's College Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DUNNS-AFPFY112-RFUMA
Record Dates: First submitted 2013-09-11; First posted 2013-09-16 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Medical; Abortion, Fetus
Keywords: medical abortion; telephone follow-up; ultrasound; serum hCG; methotrexate; misoprostol
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Follow-up (SFU) (Active Comparator): Women selecting SFU at either site (BCBC or CIHC) will schedule their in-person follow-up appointment before leaving the BCBC clinic on Study Day 1, when they receive their medication. In-person follow-up appointment will be scheduled for Study Day 15 (± 3 days)where, as per usual care, includes a history and a Post-abortion Checklist, transvaginal ultrasound, and a bimanual exam to confirm successful pregnancy expulsion.
  Interventions: Other: Standard Follow-up (SFU)
- Remote Follow-up (RFU) (Experimental): On Study Day 1 in both sites, women selecting RFU will receive 3 laboratory requisition forms for serum β-hCG testing and will be instructed to have testing done at a laboratory site of her choice on Study Day 10-12. The follow-up telephone appointment will be scheduled to take place on Study Day 15 (±3 days). For the follow-up telephone appointment, the research nurse/nurse practitioner will calculate the percentage fall in the β-hCG value. She will contact the subject by phone at the specified time, take a history of the timing of misoprostol use, resulting symptoms and complete the symptom Post-abortion Check-list. The research nurse/nurse practitioner, in consultation with the clinic physician if necessary, will confirm the information, determine whether other follow-up is required.
  Interventions: Other: Remote Follow-up (RFU)

INTERVENTIONS:
Other: Remote Follow-up (RFU) — Women in the RFU group will be asked to return to the clinic for assessment if they have any complications.
  Other Names: telephone follow-up; serum hCG
  Arms: Remote Follow-up (RFU)
Other: Standard Follow-up (SFU) — Study Day 15 (± 3 days)requires an in-person post-abortion checkup: transvaginal ultrasound, and a bimanual exam to confirm successful pregnancy expulsion.
  Other Names: In-clinic visit; Ultrasound
  Arms: Standard Follow-up (SFU)

SUMMARY:
Background: Medical abortions in Canada are provided using a standard regimen of methotrexate and misoprostol. After these medications are administered, patients are most commonly checked for termination of the pregnancy with an ultrasound and physical examination at an in-clinic follow-up appointment. These follow-up appointments can be inconvenient, costly, and take away from patient privacy. Furthermore, it has been suggested that these follow-up appointments may not be necessary for patients.

Objective: To determine whether remote follow-up, using telephone and blood testing is a feasible, safe, and effective method of follow-up after medical abortion, compared to standard care that requires an in-clinic visit and ultrasound.

This study offers women the option of remote follow-up by telephone combined with serum Beta-human chorionic gonadotropin (β-hCG) testing or standard in-clinic follow up. We will determine women's preferences for follow up, and compare adherence to the follow-up schedule, number of clinical contacts, and outcomes of the abortion. This study will be performed at two clinics in Toronto, the Bay Centre for Birth Control (BCBC) and the Choice in Health Clinic (CIHC).

Primary Hypothesis: Follow-up will be more successful with RFU, compared to SFU.

DETAILED DESCRIPTION:
The protocol is altered for women who have an ultrasound that shows only a gestational sac (no yolk sac or fetal pole). Women in both follow-up groups will have β-hCG testing on the day of methotrexate injection and again in 8 days. If the level does not fall by 50% or they have concerning symptoms, they are asked to return to clinic for evaluation. If the β-hCG level falls by 50% or more, they will continue to be followed as per the protocol in their chosen group, but will be followed until their β-hCG becomes negative.

ELIGIBILITY:
Inclusion Criteria:

1. Requests a medical abortion and fulfills standard eligibility criteria for M&M abortion:

   * Clear decision to have an abortion
   * Valid Ontario Health card
   * Willing to abstain for vaginal intercourse and alcohol for 14 days
   * Ability to insert misoprostol vaginal tablets
   * Emergency Contact number
   * Stop folic acid vitamins on initial contact
   * Good general health
   * Single intrauterine gestation less than or equal to 49 days as determined by transvaginal ultrasound
   * Telephone access
   * Access to emergency medical care within 30 minutes of home
   * Agrees to undergo a surgical abortion in case of failure of the medical abortion method
2. Ability to understand the protocol and consent
3. Willingness to comply with either the SFU or RFU follow-up schedule

Exclusion Criteria:

1. Factors that exclude women from eligibility for M&M abortion:

   * Coagulopathy or hemoglobin less than 100, White Blood Cell count < 4.0 platelet <140,000
   * Allergy to methotrexate or misoprostol
   * Presence of an intrauterine device
   * Acute or chronic renal or hepatic disease
   * Acute inflammatory bowel disease
   * Uncontrolled seizure disorder
   * Sickle cell anemia
   * Breastfeeding
   * Chronic oral corticosteroid therapy
   * Any condition that in the opinion of the clinician investigator would compromise the safety of medical abortion for this patient
2. Requires the support of an interpreter

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2011-07; Primary Completion 2013-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Rate of successful follow-up in women choosing RFU compared with those choosing SFU after medical abortion with M&M | Within the designated time of 15 days post methotrexate injection ±3 days
  Successful follow-up will be defined as completion of telephone follow-up contact and serum β-hCG testing (for the RFU cohort) or attendance for the in-clinic follow-up visit within the designated time of 15 days post methotrexate injection ±3 days (for the SFU cohort).

SECONDARY OUTCOMES:
Percent of women who choose RFU | 1 day
Percent of women choosing RFU who complete follow-up without a clinic visit | Within the designated time of 15 days post methotrexate injection ±3 days
Percent of women in RFU and SFU groups who made no unscheduled visits related to medical abortion | Within 28 days of methotrexate injection ±3 days

OTHER OUTCOMES:
Emergency department visit | Within 28 days of methotrexate injection ±3 days
  Determined through subject history
Hemorrhage - defined as bleeding resulting in transfusion, intravenous fluids or a drop in hemoglobin of 20 g | Within 28 days of methotrexate injection ±3 days
  Determined from patient history with retrieval of emergency department/hospital records or documented drop of 20 g.
D&C with the cause characterized as 1) for bleeding, at clinician's recommendation, 2) for continuing pregnancy, 3) at patient's request (usually because of delayed expulsion of the pregnancy in a medically stable patient) | Within 35 days of methotrexate injection
Infection requiring antibiotics | Within 28 days of methotrexate injection ±3 days
  Determined from the clinic record or subject history
Acceptability of SFU and RFU | At 28 days after methotrexate injection ±3 days
  Measured using an Acceptability Questionnaire administered at discharge from ongoing care. This questionnaire is adapted from a previous study of acceptability of mifepristone and misoprostol abortions by Winikoff et al. It contains four close-ended and three open-ended questions designed to capture the patient's perspective on their medical abortion experience, whether they would choose the same method of follow-up in future, and their opinions on the best and worst features of their chosen follow-up method.
Number of subject-initiated telephone contacts during clinic hours | Within 28 days of methotrexate injection ±3 days
  Abstracted from the medical record
Number of subject-initiated telephone contacts to on-call physician | Within 28 days of methotrexate injection ±3 days
  Abstracted from the medical record
Number of clinic-initiated telephone contacts outside of the scheduled follow-up contact for the RFU group | Within 28 days of methotrexate injection ±3 days
  Abstracted from the medical record
Number of letters sent | Within 28 days of methotrexate injection ±3 days
  Abstracted from the medical record
Selected method of contraception | At 28 days after methotrexate injection ±3 days
Reason for choice of follow-up method | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Dunn, MD MSc CCFP, Principal Investigator — Women's College Hospital, University of Toronto
Locations (2):
- Canada (2):
  - Women's College Hospital-Bay Center for Birth Control, Toronto, Ontario
  - Choice in Health Clinic, Toronto, Ontario

REFERENCES:
- [Background] Perriera LK, Reeves MF, Chen BA, Hohmann HL, Hayes J, Creinin MD. Feasibility of telephone follow-up after medical abortion. Contraception. 2010 Feb;81(2):143-9. doi: 10.1016/j.contraception.2009.08.008. Epub 2009 Sep 30. PMID 20103453
- [Background] Clark W, Panton T, Hann L, Gold M. Medication abortion employing routine sequential measurements of serum hCG and sonography only when indicated. Contraception. 2007 Feb;75(2):131-5. doi: 10.1016/j.contraception.2006.08.001. Epub 2006 Dec 22. PMID 17241843
- [Background] Clark W, Bracken H, Tanenhaus J, Schweikert S, Lichtenberg ES, Winikoff B. Alternatives to a routine follow-up visit for early medical abortion. Obstet Gynecol. 2010 Feb;115(2 Pt 1):264-272. doi: 10.1097/AOG.0b013e3181c996f3. PMID 20093898
- [Background] Kaneshiro B, Edelman A, Sneeringer RK, Ponce de Leon RG. Expanding medical abortion: can medical abortion be effectively provided without the routine use of ultrasound? Contraception. 2011 Mar;83(3):194-201. doi: 10.1016/j.contraception.2010.07.023. Epub 2010 Sep 17. PMID 21310279
- [Background] Fiala C, Safar P, Bygdeman M, Gemzell-Danielsson K. Verifying the effectiveness of medical abortion; ultrasound versus hCG testing. Eur J Obstet Gynecol Reprod Biol. 2003 Aug 15;109(2):190-5. doi: 10.1016/s0301-2115(03)00012-5. PMID 12860340
- [Background] Creinin MD, Vittinghoff E, Keder L, Darney PD, Tiller G. Methotrexate and misoprostol for early abortion: a multicenter trial. I. Safety and efficacy. Contraception. 1996 Jun;53(6):321-7. doi: 10.1016/0010-7824(96)00080-7. PMID 8773418
- [Background] von Hertzen H, Honkanen H, Piaggio G, Bartfai G, Erdenetungalag R, Gemzell-Danielsson K, Gopalan S, Horga M, Jerve F, Mittal S, Ngoc NT, Peregoudov A, Prasad RN, Pretnar-Darovec A, Shah RS, Song S, Tang OS, Wu SC; WHO Research Group on Post-Ovulatory Methods for Fertility Regulation. WHO multinational study of three misoprostol regimens after mifepristone for early medical abortion. I: Efficacy. BJOG. 2003 Sep;110(9):808-18. doi: 10.1111/j.1471-0528.2003.02430.x. PMID 14511962
- [Background] Schaff EA, Fielding SL, Westhoff C. Randomized trial of oral versus vaginal misoprostol at one day after mifepristone for early medical abortion. Contraception. 2001 Aug;64(2):81-5. doi: 10.1016/s0010-7824(01)00229-3. PMID 11704083
- [Background] Rossi B, Creinin MD, Meyn LA. Ability of the clinician and patient to predict the outcome of mifepristone and misoprostol medical abortion. Contraception. 2004 Oct;70(4):313-7. doi: 10.1016/j.contraception.2004.04.005. PMID 15451336